## Enhanced Virologic Monitoring for Pregnant and Postpartum Women With HIV

Study Protocol Approved July 27, 2023

# **Principal Investigators:**

Dr. James Ayieko, MBChB, MPH, PhD KEMRI - CMR

Pamela Murnane, PhD, MPH University of California, San Francisco

## **Brief Summary:**

The goal of this study is to learn about supporting pregnant and postpartum women living with HIV with treatment adherence. The investigators will conduct a pilot study of an intervention that includes peer counseling about viral load levels and rapid delivery of viral load results. The investigators will evaluate the feasibility of the intervention, and will assess whether it improves viral suppression 6 months following the intervention, compared to historical controls.

#### **Detailed Description:**

The investigators will examine the use of more frequent virologic monitoring with enhanced communication around low-level viremia as a strategy to identify and support pregnant and postpartum women at risk of virologic failure. Virologic monitoring itself can reinforce adherence in stable patients, and more frequent monitoring can detect potential adherence challenges early. Notably, low-level viremia is a strong predictor of subsequent virologic failure, and the lowest level associated with perinatal transmission is not known.

The pilot study will run for 6 months at 4 Ministry of Health facilities in Kisumu County, Kenya; 275 participants will be enrolled. Prior to the pilot study, 125 controls will be enrolled prospectively, and 150 controls will be abstracted from records from the prior year.

## 1. INTRODUCTION/BACKGROUND

Emerging estimates of virologic suppression fall far short of the UNAIDS target among pregnant and postpartum women living with HIV on antiretroviral therapy (ART) in sub-Saharan Africa. The UNAIDS 90-90-90 targets to help end the AIDS epidemic are: 90% of persons living with HIV know their status; 90% of those who know their status are on ART; 90% of those on ART are virologically suppressed. Lack of virologic suppression magnifies the risk of disease progression and sexual and perinatal transmission of the virus. The emerging estimates of viremia build on the concerning recent meta-analysis reporting 24% of pregnant women and 43% of postpartum women had suboptimal ART adherence across 51 studies, including 6 from Kenya and 5 each from South Africa and Zambia. Several studies have shown

that the vast majority of viremia experienced perinatally and otherwise is due to suboptimal adherence to ART rather than acquired resistance.<sup>5,9-11</sup> Reaching the third 90 target requires a lifelong commitment to optimal ART adherence. However, pregnancy and the postpartum period introduce significant transitions in daily routines which present both unique challenges to medication adherence and unique opportunities for intervention.

**Evidence-based strategies to improve adherence and reduce viremia risk are not always optimally delivered to pregnant and postpartum women most in need of support.** For persons with or "at risk" of virologic failure, Kenyan guidelines are in place for enhanced virologic monitoring, enhanced adherence assessment and counseling, and enhanced referrals for nutrition and psychosocial support. However, strategies are needed to identify persons "at risk" of virologic failure, prior to detection of viremia or at the earliest possible time-point of non-suppression, to optimize delivery of timely enhanced support. Such services provided after virologic failure occurs may come too late to prevent the development of resistance or transmission of the virus.

Virologic monitoring can reinforce adherence in stable patients. With frequent monitoring, adherence challenges can be detected and addressed early. In addition, low-level viremia is a strong predictor of subsequent failure, and the level associated with perinatal transmission is not known. Thus, using a sensitive viral load assay (lower limit of detection ≤100 copies/mL) every 3 months in pregnancy and up to 6 months postpartum could provide an opportunity to provide enhanced support early.

The scientific premise of this proposal is that enhanced virologic monitoring has the potential to improve health outcomes in the highest risk patients. Early adherence support for pregnant and postpartum women most at risk of viremia could have an important impact on reaching the UNAIDS third 90 target in this population, and ultimately on improved maternal and infant outcomes among women living with HIV.

## 2. OBJECTIVES

**Objective**: Evaluate the implementation and potential impact of risk assessment with enhanced virologic monitoring to facilitate targeted, evidence-based adherence support to pregnant/postpartum women at risk of viremia in a pilot study in western Kenya.

# 3. <u>DESIGN AND METHODOLOGY</u>

The study will be conducted within MoH clinics, in Kisumu County, Kenya. Kisumu County is one of the regions of Kenya most affected by the HIV epidemic: in 2015, adult HIV prevalence (age 15-49) was 20% and the rate of perinatal transmission was 20%.<sup>48</sup>

In a 6-month pilot study, we will evaluate the implementation and potential impact of enhanced virologic monitoring for pregnant and postpartum women living with HIV to reduce the risk of viremia and loss from care. Prior to the pilot study, we will sample 2 control groups: 1) 125 women will be prospectively enrolled at the pilot study sites (as part of the CAPS mobility substudy), and 2) 150-320 women will be randomly selected from de-identified electronic medical records.

- (a) Study sites: 2-4 clinics will be selected for the pilot study.
- **(b) Study populations**: All women seeking care at these sites who are on ART *and*, either in their 3<sup>rd</sup> trimester of pregnancy, in the maternity ward for delivery, or within the first 6 months postpartum are eligible. Our rationale for this time range is: (1) Late pregnancy and delivery are critical periods for prevention of mother to child transmission. (2) 0-6 months postpartum is a period highly susceptible to disengagement from care among women living with HIV.
- **(c) Sampling**: For prospectively enrolled controls and pilot study participants, to ensure adequate representation from each facility and to avoid seasonal differences by site, we will conduct recruitment at each site simultaneously, visiting each site within any given week in which recruitment is done, to the best our ability. We will invite all women attending clinic on days of recruitment at each site, and will trace all women late for visits that were due on those recruitment days. Controls selected from records only will be randomly sampled from eligible women with viral loads scheduled for collection in the 6 months prior to the pilot study.

## Recruitment.

Building on our established relationships with MoH and clinic leadership in Kisumu, we will work collaboratively with these teams to ensure on-site research staff support with patient recruitment, including access to patients, clinic records, and registers. We will attempt to recruit, consent, enroll, and conduct baseline visits in conjunction with a clinic visit to reduce the burden on participants. For participants that prefer to meet elsewhere, we will arrange a separate time and place to meet at their convenience. For those who are late for visits, mentor mothers will use all available phone numbers and location data in the clinical record to locate the individual. For participants who are hard to reach, we will train mentor mothers with established tracking methods to determine potential relocation information about the participant.<sup>51</sup>

#### (d) Procedures:

## Study visit

For prospectively enrolled controls and pilot study participants, following participant consent, study staff/providers will collect sociodemographic, clinical, and mobility questionnaires from patients directly and from records, and a blood sample to test viral load. Study staff/providers will have access to clinical records during the study visit and can query patients and clinical staff regarding key clinical variables if data are missing from records. Sociodemographic data and mobility measures will be collected directly from the participant. Data will be collected directly into REDCap, a secure platform for building and managing datasets which has an off-line data collection option enabling use in settings where internet access may be limited.

For participants who are reached and consented outside of the clinic via tracing, data will be collected in a location convenient to the patient.

Samples collected for viral load testing will immediately be stored in a cooler bag and will be tested for HIV RNA levels with Cephied's GeneXpert® technology, Xpert HIV-1 Viral Load on the same day.

## Intervention

Our enhanced virologic monitoring intervention includes 3 components: 1) More frequent viral load collection than standard of care, 2) Rapid return of viral load results, 3) Enhanced viral load counselling, including about low-level viremia. These are detailed below.

## 1) More frequent viral load collection

Our research assistants will be trained in phlebotomy. All participants who have not had a viral load collected within the prior 80 days will have a blood sample collected at baseline for viral load testing. Those who enroll in the first 3 months of the pilot study period will be eligible for a follow-up visit within the 6-month pilot study period, and will have viral load assessed again at the 3-month follow up visit.

## 2) Rapid return of viral load results:

Mentor mothers will be trained to return viral load results to patients with scripted messaging according to viral load level (undetectable, low-level viremia (50-1000), high viral load (>1000)). Patients will be offered a choice of the mode of delivery, including text, phone, or in-person. Detectable viral loads will not be delivered by text, and women with high viral loads may be asked to return to the clinic for in-person counselling.

#### 3) Enhanced viral load counselling

Mentor mothers will reinforce adherence with all patients with undetectable levels via scripted messaging to reward and encourage healthy behavior. For those with any detectable levels, mentor mothers will be trained to provide targeted counseling about low-level and higher viral loads. Women who report significant psychosocial barriers will be referred to a social worker.

## Study Measures.

## Baseline characteristics.

To assess objective 3 and the objectives of the sub-study, we will collect information about women's baseline characteristics (individual and social) that we believe may be confounders of the associations we plan to estimate (ie., the impact of enhanced virologic monitoring on subsequent viremia; the impact of mobility on viremia and retention in care). These baseline characteristics will include the following, and the surveys are included as an appendix to this protocol:

- Sociodemographic and health information (e.g., marital status, education, mobility)
- Clinical records data abstraction (pregnancy history, HIV history from records)
- Household food insecurity scale (HFIAS)
- Perceived stress scale (to measure psychosocial stress)
- Edinburgh depression scale (to measure perinatal depression)

If, during the depression questionnaire, a study participant expresses an intent to harm themselves or scores 11 or higher,<sup>52</sup> they will be referred to social services (e.g., social worker, psychiatrist, other mental health provider) for further assessment on the same day. Because this questionnaire will be collected on REDCap, the score will be automatically generated once the form is completed. The social service staff member is not part of the study team. The study will cover the cost of an initial consultation for patients who would benefit from further assessment up to ~2000 KShs or ~\$20 USD. If further care is recommended, the participant will be responsible for those costs. We note these potential costs in the informed consent form.

#### HIV care outcomes.

The viral loads collected as part of the intervention will guide the counselling that is provided during the study. Study outcome viral loads will be routine care viral loads that are collected (1) within the 6 months following the control participants enrollment (and only) study visit, for prospectively enrolled controls, (2) within the 6 months prior to the pilot study for controls

retrieved from electronic records, and (3) within the 6 months following the pilot participants last study visit. The study team will work together with the clinical teams to ensure these viral load outcomes are measured and recorded according to national guidelines. Viremia will be defined as any detectable levels of HIV RNA. <u>Suboptimal care engagement</u> will be defined as late for a clinic visit by 30 days or more.

## Implementation outcomes.

Enola Proctor has proposed a taxonomy of implementation outcomes to inform systematic and scientifically rigorous measurement of implementation success. The pilot study outcomes summarized in Table 1 are outcomes which Proctor has identified as most salient to the early stages of implementation, while gaining training in the measurement of later stage outcomes to incorporate in my future research.

Table 1. Implementation outcomes and method of measurement in the pilot study

| Outcome | Method of measurement | When measured |
|---|---|---|
| Acceptability<br>(provider satisfaction,<br>facilitators, barriers) | Survey | End of pilot |
| Adoption<br>(uptake, intention) | <ul> <li>Record for each enrolled participant</li> <li>whether the viral load monitoring was conducted on schedule</li> <li>what action was taken in response to low-level viremia</li> <li>reasons for no action</li> </ul> | Daily throughout follow-up |
| Appropriateness (perceived fit) | • Survey | End of pilot |
| Feasibility<br>(practicability, utility) | • Survey | End of pilot |

The PIs and research team will lead training sessions for mentor mothers and research assistants prior to the start of the study, followed by periodic (at least monthly) follow-up sessions to reinforce initial plans and revise strategies as needed. These data will be entered into de-identified REDCap databases containing only anonymous study IDs. A separate secure list linking study IDs to clinic IDs will be maintained in order to later link these records to virologic outcomes. At the conclusion of the study, <u>surveys</u> will be administered to key stakeholders and care providers at the sites (n=~10) to measure acceptability and feasibility, and <u>semi-structured in-depth interviews</u> will be conducted to further assess acceptability, appropriateness and intentions. Interview guides will be informed by a rapid analysis of survey data and assessments of adoption.

<u>Evaluating the potential impact on maternal viremia</u>. We acknowledge that this pre-post analysis will not reflect a causal effect of the pilot on viremia risk, as any observed differences could be due to temporal or other factors. This pilot study, rather, aims to explore the *potential* impact while gathering critical data on the feasibility and acceptability of the intervention to inform future research.

## 4. DATA MANAGEMENT

<u>Analyses of implementation outcomes</u>. Analyses will summarize acceptability and feasibility survey results, summaries of adoption, as well as the clinical and sociodemographic characteristics of the women seen at the clinic during the pilot study, using descriptive statistics.

<u>Evaluating the potential impact on maternal viremia</u>. The frequency of viremia in the year preceding the pilot to the frequency among women seeking care during the pilot will be

compared with logistic regression, adjusted for baseline differences in clinical and demographic characteristics.

#### 5. ETHICAL CONSIDERATIONS

Study databases will only include anonymous study IDs. In order to link baseline patient characteristics to viral load outcomes, we will maintain a separate secure list linking study IDs to clinic IDs. Only the PI and research team will have access to this linked ID list, and will use it to ensure data quality.

<u>Potential risks</u> will be minimal, and could include 1) discomfort having additional blood draws for additional viral load testing, and 2) loss of privacy or social harms due to loss of privacy.

<u>Informed consent</u>: We will obtain written informed consent from all women participating. Clinical care remains at the discretion of the treating clinician. The informed consent forms will describe the purpose of the study, the types of activities that will be conducted, and the risks and benefits of participation.

Protections Against Risk: Every effort will be made to ensure the privacy of participants. All study paper and study databases will only include de-identified data and study IDs. Lists matching study IDs to clinic IDs and provider names will be maintained in a separate REDCap project only accessible to the PI and the research assistant. Recording devices and paper informed consent forms, interview and observation notes, and any other paper materials containing human subject data will be stored in a locked file cabinet in a locked room. Audio recordings and interview transcripts will be stored in secure, password-protected, MyResearch online storage space to allow access in Kenya and San Francisco. MyResearch is supported in a secure, professional data center, locked and quarded 24x7 with UCSF badge access required for physical entry. Data exists on a private network with its own firewall. REDCap is housed in a locked and guarded data center. Entrance to the data center requires triple factor authentication: use of a card key to unlock the data center door, biometric authentication and a second card key lock secures the cage that the servers reside within. The security of the data center is monitored by a security camera system. REDCap servers are guarded by multiple firewall and intrusion detection systems. All electronic connections to the REDCap environment are encrypted.

# 6. <u>REFERENCES</u>

- 1. Myer L, Dunning L, Lesosky M, Hsiao NY, Phillips T, Petro G, et al. Frequency of viremic episodes in HIV-infected women initiating antiretroviral therapy during pregnancy: a cohort study. Clinical Infectious Diseases. 2017;64(4):422-7. Epub 2016/12/09.
- 2. Chetty T, Newell ML, Thorne C, Coutsoudis A. Viraemia before, during and after pregnancy in HIV-infected women on antiretroviral therapy in rural KwaZulu-Natal-South Africa, 2010-2015. Tropical Medicine and International Health, 2017, Epub 2017/11/10.
- 3. Hoffman RM, Warshaw M, Amico KR, Pilotto J, Masheto G, Achalapong J, et al. Predictors of virologic failure in postpartum women on ART in PROMISE 1077HS. Conference on Retroviruses and Opportunistic Infections; Mar 4-7; Boston, MA. 2018.
- 4. Odayar J, Abrams EJ, Zerbe A, Phillips TK, Myer L. Early clinical events after ART initiation in pregnancy influence viral load outcomes. Conference on Retroviruses and Opportunistic Infections; Mar 4-7; Boston, MA. 2018.

- 5. Currier JS, Britto P, Hoffman RM, Brummel S, Masheto G, Joao E, et al. Randomized trial of stopping or continuing ART among postpartum women with pre-ART CD4 >/= 400 cells/mm3. PloS One. 2017;12(5):e0176009. Epub 2017/05/11. PMCID: PMC5425014.
- 6. Ronen K, Khasimwa B, Chohan B, Matemo D, Unger J, Drake AL, et al. Disparities in antenatal virologic failure among women receiving Option B+ in Kenya. Conference on Retroviruses and Opportunistic Infections; Mar 4-7; Boston, MA. 2018.
- 7. UNAIDS. 90-90-90 An ambitious treatment target to help end the AIDS epidemic. Geneva, Switzerland: 2014.
- 8. Nachega JB, Uthman OA, Anderson J, Peltzer K, Wampold S, Cotton MF, et al. Adherence to antiretroviral therapy during and after pregnancy in low-income, middle-income, and high-income countries: a systematic review and meta-analysis. AIDS. 2012;26(16):2039-52. PMCID: PMC5061936.
- 9. Hosseinipour M, Nelson JAE, Trapence C, Rutstein SE, Kasende F, Kayoyo V, et al. Viral suppression and HIV drug resistance at 6 months among women in Malawi's Option B+ Program: results from the PURE Malawi Study. Journal of Acquired Immune Deficiency Syndromes. 2017;75 Suppl 2:S149-S55. Epub 2017/05/13. PMCID: PMC5431274.
- 10. Ruperez M, Noguera-Julian M, Gonzalez R, Maculuve S, Bellido R, Vala A, et al. HIV drug resistance patterns in pregnant women using next generation sequence in Mozambique. PloS One. 2018;13(5):e0196451. Epub 2018/05/10. PMCID: PMC5942837.
- 11. Myer L, Redd AD, Mukonda E, Lynch B, Phillips TK, Eisenberg A, et al. ART detection and resistance during viraemic episodes in pregnancy and breastfeeding. Conference on Retroviruses and Opportunistic Infections; Mar 4-7; Boston, MA. 2018.
- 12. Ministry of Health. Guidelines on Use of Antiretroviral Drugs for Treating and Preventing HIV Infection in Kenya. 2016.
- 13. Sheridan SL, Crespo E. Does the routine use of global coronary heart disease risk scores translate into clinical benefits or harms? A systematic review of the literature. BMC Health Services Research. 2008;8:60. Epub 2008/03/28. PMCID: PMC2294118.
- 14. Sosenko JM, Skyler JS, Palmer JP, Diabetes Type T, Diabetes Prevention Trial-Type 1 Study G. The development, validation, and utility of the Diabetes Prevention Trial-Type 1 Risk Score (DPTRS). Current Diabetes Reports. 2015;15(8):49. Epub 2015/06/17. PMCID: PMC4795007.
- 15. Long B, Long D, Koyfman A. Emergency medicine evaluation of community-acquired pneumonia: history, examination, imaging and laboratory assessment, and risk scores. Journal of Emergency Medicine. 2017;53(5):642-52. Epub 2017/09/25.
- 16. Koss CA, Ayieko J, Mwangwa F, Owaraganise A, Kwarisiima D, Balzer LB, et al. Early Adopters of HIV Preexposure Prophylaxis in a Population-based Combination Prevention Study in Rural Kenya and Uganda. Clinical Infectious Diseases. 2018. Epub 2018/05/10.
- 17. Irungu EM, Heffron R, Mugo N, Ngure K, Katabira E, Bulya N, et al. Use of a risk scoring tool to identify higher-risk HIV-1 serodiscordant couples for an antiretroviral-based HIV-1 prevention intervention. BMC Infectious Diseases. 2016;16(1):571. Epub 2016/10/19. PMCID: PMC5067880.
- 18. Mungwira RG, Divala TH, Nyirenda OM, Kanjala M, Muwalo F, Mkandawire FA, et al. A targeted approach for routine viral load monitoring in Malawian adults on antiretroviral therapy. Tropical Medicine and International Health. 2018;23(5):526-32. Epub 2018/03/06. PMCID: PMC5932246.
- 19. Phan V, Thai S, Koole O, Menten J, Meheus F, van Griensven J, et al. Validation of a clinical prediction score to target viral load testing in adults with suspected first-line

- treatment failure in resource-constrained settings. Journal of Acquired Immune Deficiency Syndromes. 2013;62(5):509-16. Epub 2013/01/22.
- 20. van Griensven J, Phan V, Thai S, Koole O, Lynen L. Simplified clinical prediction scores to target viral load testing in adults with suspected first line treatment failure in Phnom Penh, Cambodia. PloS One. 2014;9(2):e87879. Epub 2014/02/08. PMCID: PMC3913697.
- 21. Meya D, Spacek LA, Tibenderana H, John L, Namugga I, Magero S, et al. Development and evaluation of a clinical algorithm to monitor patients on antiretrovirals in resource-limited settings using adherence, clinical and CD4 cell count criteria. Journal of the International AIDS Society. 2009;12:3. Epub 2009/03/06. PMCID: PMC2664320.
- 22. Petersen ML, LeDell E, Schwab J, Sarovar V, Gross R, Reynolds N, et al. Super Learner analysis of electronic adherence data improves viral prediction and may provide strategies for selective HIV RNA monitoring. Journal of Acquired Immune Deficiency Syndromes. 2015;69(1):109-18. Epub 2015/05/06. PMCID: PMC4421909.
- 23. Robbins GK, Johnson KL, Chang Y, Jackson KE, Sax PE, Meigs JB, et al. Predicting virologic failure in an HIV clinic. Clinical Infectious Diseases. 2010;50(5):779-86. Epub 2010/02/04. PMCID: PMC3101804.
- 24. Steyerberg EW, Moons KG, van der Windt DA, Hayden JA, Perel P, Schroter S, et al. Prognosis Research Strategy (PROGRESS) 3: prognostic model research. PLoS Medicine. 2013;10(2):e1001381. Epub 2013/02/09. PMCID: PMC3564751.
- 25. Taylor BS, Garduno LS, Reyes EV, Valino R, Rojas R, Donastorg Y, et al. HIV care for geographically mobile populations. Mount Sinai Journal of Medicine. 2011;78(3):342-51. PMCID: PMC3100665.
- 26. Andrews JR, Wood R, Bekker LG, Middelkoop K, Walensky RP. Projecting the benefits of antiretroviral therapy for HIV prevention: the impact of population mobility and linkage to care. Journal of Infectious Diseases. 2012;206(4):543-51. PMCID: PMC3491737.
- 27. Taylor BS, Reyes E, Levine EA, Khan SZ, Garduno LS, Donastorg Y, et al. Patterns of geographic mobility predict barriers to engagement in HIV care and antiretroviral treatment adherence. AIDS Patient Care and STDS. 2014;28(6):284-95. PMCID: PMC4046197.
- 28. Marson KG, Tapia K, Kohler P, McGrath CJ, John-Stewart GC, Richardson BA, et al. Male, mobile, and moneyed: loss to follow-up vs. transfer of care in an urban African antiretroviral treatment clinic. PloS One. 2013;8(10):e78900. Epub 2013/11/10. PMCID: PMC3812001.
- 29. Ayieko J, Charlebois ED, Getahun M, Maeri I, Eyul P, Murnane PM, et al. Challenges to HIV care engagement among mobile populations in rural Kenya and Uganda. Conference on Retroviruses and Opportunistic Infections Mar 8-11; Boston, MA 2020.
- 30. Bernardo EL, Nhampossa T, Clouse K, Carlucci JG, Fernandez-Luis S, Fuente-Soro L, et al. Patterns of mobility and its impact on retention in care among people living with HIV in the Manhica District, Mozambique. PloS One. 2021;16(5):e0250844. Epub 2021/05/22. PMCID: PMC8139482.
- 31. Deshingkar P, Grimm S. Internal Migration and Development: A Global Perspective. Geneva, Switzerland: 2005.
- 32. Phillips TK, Clouse K, Zerbe A, Orrell C, Abrams EJ, Myer L. Linkage to care, mobility and retention of HIV-positive postpartum women in antiretroviral therapy services in South Africa. Journal of the International AIDS Society. 2018;21 Suppl 4:e25114. Epub 2018/07/22. PMCID: PMC6053482.
- 33. Clouse K, Vermund SH, Maskew M, Lurie MN, MacLeod W, Malete G, et al. Mobility and Clinic Switching Among Postpartum Women Considered Lost to HIV Care in South Africa. Journal of Acquired Immune Deficiency Syndromes. 2017;74(4):383-9. PMCID: PMC5324708.

- 34. Clouse K, Fox MP, Mongwenyana C, Motlhatlhedi M, Buthelezi S, Bokaba D, et al. "I will leave the baby with my mother": Long-distance travel and follow-up care among HIV-positive pregnant and postpartum women in South Africa. Journal of the International AIDS Society. 2018;21 Suppl 4:e25121. Epub 2018/07/22. PMCID: PMC6053484.
- 35. Ssetaala A, Ssempiira J, Nanyonjo G, Okech B, Chinyenze K, Bagaya B, et al. Mobility for maternal health among women in hard-to-reach fishing communities on Lake Victoria, Uganda; a community-based cross-sectional survey. BMC Health Services Research. 2021;21(1):948. Epub 2021/09/11. PMCID: PMC8431852.
- 36. Ferguson L, Lewis J, Grant AD, Watson-Jones D, Vusha S, Ong'ech JO, et al. Patient attrition between diagnosis with HIV in pregnancy-related services and long-term HIV care and treatment services in Kenya: a retrospective study. Journal of Acquired Immune Deficiency Syndromes. 2012;60(3):e90-7.
- 37. Deane KD, Parkhurst JO, Johnston D. Linking migration, mobility and HIV. Tropical Medicine and International Health. 2010;15(12):1458-63.
- 38. Murnane PM, Gandhi M, Bacchetti P, Getahun M, Gutin SA, Okochi H, et al. Distinct forms of migration and mobility are differentially associated with HIV treatment adherence. AIDS. 2022; In press.
- 39. World Health Organization. Consolidated guideline on the use of antiretroviral drugs for treating and preventing HIV infection: recommendations for a public health approach. Geneva, Switzerland: World Health Organization, 2016.
- 40. Office of the U.S. Global AIDS Coordinator. PEPFAR 3.0. Controlling the epidemic: delivering on the promise of an AIDS-free generation. 2014.
- 41. International AIDS Society, World Health Organization, United States President's Emergency Plan for AIDS Relief, Centers for Disease Control and Prevention, United States Agency for International Development, Global Fund to Fight AIDS Tuberculosis and Malaria, et al. Differentiated Service Delivery 2018 [cited 2018 August 2]. Available from: <a href="http://www.differentiatedservicedelivery.org/">http://www.differentiatedservicedelivery.org/</a>.
- 42. McNairy ML, Abrams EJ, Rabkin M, El-Sadr WM. Clinical decision tools are needed to identify HIV-positive patients at high risk for poor outcomes after initiation of antiretroviral therapy. PLoS Medicine. 2017;14(4):e1002278. Epub 2017/04/19. PMCID: PMC5395167.
- 43. Myer L, Essajee S, Broyles LN, Watts DH, Lesosky M, El-Sadr WM, et al. Pregnant and breastfeeding women: A priority population for HIV viral load monitoring. PLoS Medicine. 2017;14(8):e1002375. Epub 2017/08/16. PMCID: PMC5557351.
- 44. Fowler MG, Qin M, Fiscus SA, Currier JS, Flynn PM, Chipato T, et al. Benefits and risks of antiretroviral therapy for perinatal HIV prevention. New England Journal of Medicine. 2016;375(18):1726-37. PMCID: PMC5214343.
- 45. Flynn PM, Taha TE, Cababasay M, Fowler MG, Mofenson LM, Owor M, et al. Prevention of HIV-1 transmission through breastfeeding: efficacy and safety of maternal antiretroviral therapy versus infant nevirapine prophylaxis for duration of breastfeeding in HIV-1-infected women with high CD4 cell count (IMPAACT PROMISE): A randomized, open-label, clinical trial. Journal of Acquired Immune Deficiency Syndromes. 2018;77(4):383-92. Epub 2017/12/15. PMCID: PMC5825265.
- 46. Taha TE, Brummel S, Angelidou K, Fowler MG, Flynn PM, Mukuzunga C, et al. PROMISE trial: results of continued vs discontinued ART after end of breastfeeding. Conference on Retroviruses and Opportunistic Infections; Mar 4-7; Boston, MA. 2018.
- 47. Widen EM, Tsai I, Collins SM, Wekesa P, China J, Krumdieck N, et al. HIV infection and increased food insecurity are associated with adverse body composition changes among pregnant and lactating Kenyan women. European Journal of Clinical Nutrition. 2018. Epub 2018/09/07.

- 48. Ministry of Health, National AIDS Control Council. Kenya AIDS Response Progress Report 2016. Nairobi, Kenya: 2016.
- 49. Green LW. Toward cost-benefit evaluations of health education: some concepts, methods, and examples. Health Education and Behavior. 1974;2(1):34-64.
- 50. Bernard HR. Research methods in anthropology: qualitative and quantitative approaches. 5th ed. Lanhan, MD: AltaMira; 2011.
- 51. Geng EH, Glidden DV, Emenyonu N, Musinguzi N, Bwana MB, Neilands TB, et al. Tracking a sample of patients lost to follow-up has a major impact on understanding determinants of survival in HIV-infected patients on antiretroviral therapy in Africa. Tropical Medicine and International Health. 2010;15 Suppl 1:63-9. PMCID: PMC3038920.
- 52. Levis B, Negeri Z, Sun Y, Benedetti A, Thombs BD, Group DESDE. Accuracy of the Edinburgh Postnatal Depression Scale (EPDS) for screening to detect major depression among pregnant and postpartum women: systematic review and meta-analysis of individual participant data. BMJ. 2020;371:m4022. Epub 2020/11/13. PMCID: PMC7656313 at www.icmje.org/coi disclosure.pdf and declare: support from Canadian Institutes of Health Research for the submitted work; no financial relationships with any organisations that might have an interest in the submitted work in the previous three years with the following exceptions: MTo declares that he has received a grant from Merck Canada, outside the submitted work; SNV declares that she receives royalties from UpToDate, outside the submitted work; CTB declares that she receives royalties for her Postpartum Depression Screening Scale published by Western Psychological Services; PMBo declares that he receives grants and personal fees from Servier, grants from Lundbeck, and personal fees from AstraZeneca, all outside the submitted work; LMH declares that she has received personal fees from NICE Scientific Advice, outside the submitted work; ISP declares that she has served on advisory boards and acted as invited speaker at scientific meetings for MSD, Novo Nordisk, Bayer Health Care, and Lundbeck A/S: KAY declares that she receives royalties from UpToDate, outside the submitted work. All authors declare no other relationships or activities that could appear to have influenced the submitted work. No funder had any role in the design and conduct of the study; collection, management, analysis, and interpretation of the data; preparation, review, or approval of the manuscript; and decision to submit the manuscript for publication.
- 53. Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, et al. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Administration and Policy in Mental Health. 2011;38(2):65-76. Epub 2010/10/20. PMCID: PMC3068522.
- 54. Creswell JW. Data Collection. Qualitative inquiry and research design Thousand Oaks, CA: SAGE Publications; 2013. p. 145-78.
- 55. Tibshirani R. Regression shrinkage and selection via the lasso. Journal of the Royal Statistical Society Series B (Methodological). 1996;58(1):267-88.
- van der Laan MJ, Polley EC, Hubbard AE. Super learner. Statistical Applications in Genetics and Molecular Biology. 2007;6:Article25. Epub 2007/10/04.
- 57. Harrell FE, Jr., Lee KL, Mark DB. Multivariable prognostic models: issues in developing models, evaluating assumptions and adequacy, and measuring and reducing errors. Statistics in Medicine. 1996;15(4):361-87. Epub 1996/02/28.
- 58. Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Medical Care. 2012;50(3):217-26. Epub 2012/02/09. PMCID: PMC3731143.